CLINICAL TRIAL: NCT06377046
Title: Accelerated PACing for Improved Quality of lifE in Symptomatic Atrial Fibrillation Patients Undergoing Pace-and-ablate Strategy With Left Bundle Branch Area Pacing: a Randomized Controlled Pilot Trial: PACE-AF
Brief Title: Accelerated Pacing in Patients Undergoing Pace-and-ablate Strategy With LBBAP: a Randomized Controlled Pilot Trial
Acronym: PACE-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL86643.068.24
Record Dates: First submitted 2024-03-20; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Permanent Atrial Fibrillation; Persistent Atrial Fibrillation; Pacemaker DDD; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Randomized, single center, prospective, single blinded, parallel group, pilot-trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated pacing (lower rate pacemaker 80bpm) (Experimental): Patients in the experimental arm will have their pacemaker programmed to a lower rate of 80bpm.
  Interventions: Device: Accelerated pacing
- Current standard of care (lower rate pacemaker 60bpm) (Active Comparator): Patients in the control arm will have their pacemaker programmed to a lower rate of 60bpm, which is the current standard of care.
  Interventions: Device: Current standard of care

INTERVENTIONS:
Device: Accelerated pacing — The lower rate of the pacemaker will be programmed to 80 bpm in DDDR mode with mode switch to DDIR mode.
  Arms: Accelerated pacing (lower rate pacemaker 80bpm)
Device: Current standard of care — The lower rate of the pacemaker will be programmed to the current standard of care which is 60 bpm in DDDR mode with mode switch to DDIR mode.
  Arms: Current standard of care (lower rate pacemaker 60bpm)

SUMMARY:
The goal of this clinical trial is to determine the effect of accelerated pacing (pacemaker lower rate programmed to 80bpm) compared to pacing at the standard programmed lower rate of 60bpm in symptomatic atrial fibrillation patients undergoing pace-and-ablate strategy with LBBAP.

The main question it aims to answer is:

- To determine the effect of accelerated pacing on health-related quality of life compared to the current standard of care.

Secondary questions it aims to answer are:

* To study the acute hemodynamic effect of different (accelerated) pacing rates on pulmonary capillary wedge pressure, cardiac output and arterial blood pressure among atrial fibrillation patients undergoing pace-and-ablate strategy.
* To study the long-term effects (at 6 months) of accelerated pacing compared to the current standard of care among atrial fibrillation patients undergoing pace-and-ablate strategy on:
* NT pro BNP levels
* device detected atrial fibrillation burden and daily activity
* echocardiographic measurements (LVEF, left ventricular ejection fraction; LVEDD, left ventricular end- diastolic diameter; LVESD, left ventricular end-systolic diameter; LAVI left atrial volume index; diastolic parameters; strain

DETAILED DESCRIPTION:
Rationale:

Permanent pacemaker implantation combined with atrioventricular node ablation (AVNA) reduces symptoms and improves health-related quality of life (HRQoL) in patients with symptomatic atrial fibrillation (AF). A high percentage of conventional right ventricular pacing increases the risk for pacing-induced cardiomyopathy, a risk which is presumably minimised by a form of conduction system pacing, termed left bundle branch area pacing (LBBAP). LBBAP attempts to recreate the normal physiologic activation of the heart through stimulation of the heart's own natural conduction system, thereby maintaining ventricular synchrony. This strategy may be particularly important in patients with heart failure with preserved ejection fraction (HFpEF), a diagnosis that frequently coexists with AF. The long-term programming of a patient undergoing a "pace-and-ablate strategy" (pacemaker implantation and AVNA), is such that the lower rate of the pacemaker is routinely set to 60 bpm. Previous studies have shown that accelerated pacing (ie. programming the pacemaker to a lower rate of 80bpm) may improve HRQoL in a subset of patients with HFpEF. It is therefore hypothesized that accelerated pacing will improve HRQoL in patients with symptomatic AF undergoing a pace and ablate strategy, when compared to pacing at 60 bpm, which is standard of care.

Objective:

Primary objective: To determine the effect of accelerated pacing (lower programmed rate of 80 bpm) compared to pacing at the standard programmed rate of 60 bpm on HRQoL in symptomatic AF patients undergoing pace-and-ablate strategy with LBBAP.

Secondary objectives:

* To study, in a subset of participants who give informed consent, the acute hemodynamic effect of accelerated pacing rates on pulmonary capillary wedge pressure (PCWP), cardiac output and arterial blood pressure, among AF patients undergoing a pace-and-ablate strategy with LBBAP.
* To study the long-term (6 months) effects of accelerated pacing among AF patients undergoing a pace-and-ablate strategy with LBBAP by measuring NT-proBNP levels, device detected AF-burden and daily activity, by evaluating HRQoL questionnaires (SF-36), and by assessing echocardiographic measurements (LVEF, left ventricular ejection fraction; LVEDD, left ventricular end-diastolic diameter; LVESD, left ventricular end-systolic diameter; LAVI left atrial volume index; diastolic parameters; strain) compared to pacing at the standard of care lower rate of 60bpm.
* To investigate whether participants experience symptoms of accelerated pacing (such as palpitations), based on the Atrial Fibrillation Effect on Quality-of-life (AFEQT) questionnaire, compared to standard of care.

Study design:

Randomized, single center, prospective, single blinded, parallel group, pilot-trial.

Study population:

Patients ≥ 18 years with symptomatic AF undergoing pace-and-ablate strategy.

Intervention:

- 1:1 randomization to a lower rate of DDDR 80 bpm (intervention) or a lower rate of DDDR 60 bpm (control). Duration of the study is 6 months.

In a subset of participants:

- Right heart catheterisation and invasive blood pressure measurements will be conducted to evaluate acute hemodynamic effects of different (accelerated) ventricular pacing rates during the standard of care AV node ablation.

Main study parameters/endpoints:

Primary endpoint:

Difference in HRQoL between a lower rate of 80 bpm and a lower rate of 60 bpm, based on the Minnesota Living with Heart Failure Questionnaire (MLHFQ), determined at 6 months follow-up.

Secondary endpoints:

* The acute hemodynamic effects of (accelerated) pacing at time of AVNA:

  * Pulmonary Capillary Wedge Pressure (PCWP)
  * Cardiac Output (CO)
  * Systemic arterial blood pressure
* The long-term effect of accelerated pacing on:

  * HRQoL, based on the MLHFQ and SF-36 questionnaires.
  * NT-proBNP levels
  * Device detected AF burden
  * Device detected daily activity comparing accelerated- vs control rate
  * Echocardiographic measurements (LVEF, LVEDD, LVESD, LAVI, LA strain)
* Symptoms experienced as a result of (accelerated) pacing based on the AFEQT questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Referred for pace-and-ablate strategy with LBBAP for symptomatic AF
* Left ventricular ejection fraction ≥ 40%.
* Willingness to participate, to understand the instructions and fill out the questionnaires, and ability to sign informed consent.

Exclusion Criteria:

* Infiltrative or constrictive cardiomyopathy (cardiac amyloidosis/sarcoidosis/ constrictive pericarditis)
* Severe Valvular heart disease (more than moderate valvular stenosis or regurgitation, aortic or mitral valve replacement)
* Patient participating in another interventional clinical trial
* Recent (< 3 months) Myocardial infarction (MI), Transient Ischemic Attack or Cerebro- Vascular Accident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The effect of accelerated pacing (lower programmed rate of 80 bpm) compared to pacing at the standard programmed rate of 60 bpm on health-related quality of life (HRQoL) in symptomatic AF patients undergoing pace-and-ablate strategy with LBBAP. | 6 months after the AV node ablation
  The primary endpoint of this study is the difference in HRQoL, measured with the Minnesota Living with Heart Failure Questionnaire (MLHFQ), between patients programmed to accelerated pacing with a lower rate of 80 bpm (intervention) compared to current standard of care with a lower rate of 60 bpm (control). The score in the MLHFQ can range between 0 to 105, with higher scores indicating more significant impairment in health-related quality of life.

SECONDARY OUTCOMES:
The acute hemodynamic effects of different (accelerated) pacing rates on pulmonary capillary wedge pressure (PCWP). | At the AV node ablation
  The acute effect of various accelerated pacing rates on PCWP measured by a right heart catheterization during the AV node ablation procedure among AF patients undergoing a pace-and-ablate strategy with LBBAP.
The acute hemodynamic effects of different (accelerated) pacing rates on cardiac output (CO). | At the AV node ablation
  The acute effect of various accelerated pacing rates on CO measured by a right heart catheterization during the AV node ablation procedure among AF patients undergoing a pace-and-ablate strategy with LBBAP.
The acute hemodynamic effects of different (accelerated) pacing rates on arterial blood pressure. | At the AV node ablation
  The acute effect of various accelerated pacing rates on arterial blood pressure measured invasively in the femoral artery during the AV node ablation procedure among AF patients undergoing a pace-and-ablate strategy with LBBAP.
The long-term effects of accelerated pacing on health-related quality of life based on the 36-item short form health survey (SF-36) among AF patients undergoing pace-and-ablate strategy. | 6 months after the AV node ablation
  The long-term (6 months) effects of accelerated pacing on HRQoL measured by the SF-36 questionnaire.
The long-term effects of accelerated pacing on NTproBNP levels among AF patients undergoing pace-and-ablate strategy. | 6 months after the AV node ablation
  The long-term (6 months) effects of accelerated pacing on NTproBNP levels.
The long-term effects of accelerated pacing on device detected AF burden among AF patients undergoing pace-and-ablate strategy. | 6 months after the AV node ablation
  The long-term (6 months) effects of accelerated pacing on device detected AF burden.
The long-term effects of accelerated pacing on device detected daily activity among AF patients undergoing pace-and-ablate strategy. | 6 months after the AV node ablation
  The long-term (6 months) effects of accelerated pacing on device detected daily activity.
The long-term effects of accelerated pacing on echocardiographic changes among AF patients undergoing pace-and-ablate strategy. | 6 months after the AV node ablation
  The long-term (6 months) effects of accelerated pacing on LVEF.
The long-term effects of accelerated pacing on echocardiographic changes among AF patients undergoing pace-and-ablate strategy. | 6 months after the AV node ablation
  The long-term (6 months) effects of accelerated pacing on LVEDD.
The long-term effects of accelerated pacing on echocardiographic changes among AF patients undergoing pace-and-ablate strategy. | 6 months after the AV node ablation
  The long-term (6 months) effects of accelerated pacing on LVESD.
The long-term effects of accelerated pacing on echocardiographic changes among AF patients undergoing pace-and-ablate strategy. | 6 months after the AV node ablation
  The long-term (6 months) effects of accelerated pacing on LAVI.
The long-term effects of accelerated pacing on echocardiographic changes among AF patients undergoing pace-and-ablate strategy. | 6 months after the AV node ablation
  The long-term (6 months) effects of accelerated pacing on LA-strain.
Palpitations experienced as a result of (accelerated) pacing. | 6 months after the AV node ablation
  Palpitations experienced as a result of (accelerated) pacing based on the AF effect on quality of life (AFEQT) questionnaire. Patients can score between 0 and 100, with a lower score meaning a worse outcome.

IPD SHARING:
Plan to Share IPD: Undecided